CLINICAL TRIAL: NCT01719484
Title: Functional Magnetic Resonance Imaging of Stress in Obesity
Brief Title: Functional MRI of Stress in Obesity
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 0805003899
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy: Subjects deemed to be medically healthy
- Obese: Subjects deemed to be medically obese

SUMMARY:
To examine the influence of obesity on brain activation during food cue, stress, and neutral relaxing conditions

DETAILED DESCRIPTION:
Subjects will participate in an fMRI session to examine changes in frontal and limbic brain regions with food cues, stress and neutral/relaxing imagery

ELIGIBILITY:
Inclusion Criteria:

1. Between ages 18-50 years old.
2. Able to read and write.
3. negative urine toxicology screens during intake appointments indicating no history of current or past dependence on alcohol or illicit drug use.
4. WOMEN: have a regular menstrual cycle.
5. BMI: 30 < BMI < 35 for obese subjects (upper limit of 35 selected given our experience with heavier individuals fitting comfortably in the fMRI scanner) and 18.5 < BMI <25 for normal weight subjects (Institute, 2006)

Exclusion Criteria:

1. any major neurological illness or injury and any current or prior clinically significant mental health (including PTSD) or substance use disorder (with exception of nicotine dependence) as determined by SCID interview;
2. Regular use of any psychoactive drugs including anxiolytics and antidepressants.
3. Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, liver, thyroid pathology; subjects on medications for any medical condition will be excluded.
4. Any subjects with foreign ferromagnetic metal objects in their body or other MR contraindications will be excluded including subjects who work as welders.
5. Women on oral contraceptives, peri- and post-menopausal women, and pregnant or lactating women (as alterations in stress response are associated with these states).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 obese subjects and 30 matched healthy controls will be recruited for this study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
No outcome measures for this study, this is an imaging study only | Upon study completion

CONTACTS AND LOCATIONS:
Overall Officials: Marc N Potenza, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States